CLINICAL TRIAL: NCT00301665
Title: A Phase II, Multicentre, Randomised, Double-blind, Parallel Groups, Placebo Controlled Clinical Study of Efficacy and Safety of Dysport® for Migraine Prophylaxis
Brief Title: Efficacy and Safety Study of Dysport® Used for Migraine Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-38-52120-715
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this study is to evaluate the efficacy of botulinum toxin type A (Dysport®) injections into pericranial muscles compared to placebo to prevent migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* Patients having migraine without aura or with typical aura as defined by International Headache Society criteria
* Migraine attacks have been persisting for more than 1 year
* 2 to 6 migraine attacks per month of at least moderate severity over the 3 months preceding the pre-inclusion visit
* 2 to 6 migraine attacks of at least moderate severity during the screening period

Exclusion Criteria:

* Non-migraine headaches such as tension-type headaches
* Migraine with prolonged aura, familial hemiplegic migraine, basilar migraine, migraine aura without headache, migraine with acute onset aura, ophthalmoplegic migraine, retinal migraine, complications of migraine
* Onset of migraine is after age of 50
* Overuse of acute migraine medications (individuals who take medications for acute migraine more than 10 days per month) or have a history of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2003-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Significant decrease of the number of migraine attacks with Dysport® compared to placebo. | 3 months

SECONDARY OUTCOMES:
Reduction of the intensity of the migraine attacks. | 3 months
Reduction of duration of the migraine attacks. | 3 months
Reduction of migraine medication consumption. | 3 months
Improvement of quality of life. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (9):
- Czechia (3):
  - St. Anne's Faculty Hospital, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - General Faculty Hospital, Prague
- Poland (4):
  - Medical Academy of Poznan, Poznan
  - Air Force Institute of Aviation Medicine, Warsaw
  - City Hospital of Wolomin, Wołomin
  - Voivodeship (Provincial) Specialist Hospital, Zgierz
- Slovakia (2):
  - Faculty Hospital Bratislava, Bratislava
  - Faculty Hospital, Martin